CLINICAL TRIAL: NCT02519855
Title: A Phase III, Double-Blind, Randomized, Multicenter Study to Evaluate the Immunogenicity, Safety, and Tolerability of ZOSTAVAX™ Administered Concomitantly Versus Nonconcomitantly With Quadrivalent Influenza Virus Vaccine (Inactivated)
Brief Title: Study to Evaluate Immunogenicity, Safety, and Tolerability of ZOSTAVAX™ Vaccine (Zoster Vaccine Live, V211) Administered Concomitantly Versus Nonconcomitantly With Quadrivalent Influenza Virus Vaccine (Inactivated) in Participants ≥50 Years of Age (V211-062)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-062
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Influenza Vaccines; vaxigrip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concomitant Vaccination (Experimental): ZOSTAVAX™ concomitantly with influenza vaccine on Day 1, placebo to ZOSTAVAX™ at Week 4
  Interventions: Biological: ZOSTAVAX™; Biological: Placebo to ZOSTAVAX™; Biological: Influenza Vaccine
- Nonconcomitant Vaccination (Experimental): Influenza vaccine and placebo to ZOSTAVAX™ on Day 1, ZOSTAVAX™ at Week 4
  Interventions: Biological: ZOSTAVAX™; Biological: Placebo to ZOSTAVAX™; Biological: Influenza Vaccine

INTERVENTIONS:
Biological: ZOSTAVAX™ — A single blinded administration of 0.65 mL subcutaneous injection on Day 1 (concomitant) or at Week 4 (nonconcomitant)
  Other Names: V211
Biological: Placebo to ZOSTAVAX™ — A single blinded administration of 0.65 mL subcutaneous injection on Day 1 (nonconcomitant) or at Week 4 (concomitant)
Biological: Influenza Vaccine — A single open-label administration of 0.5 mL intramuscular injection on Day 1
  Other Names: Fluzone, Vaxigrip

SUMMARY:
The study evaluated immunogenicity, safety, and tolerability of ZOSTAVAX™ Vaccine (V211) administered concomitantly versus nonconcomitantly with Quadrivalent Influenza Virus vaccine (inactivated) in participants ≥50 years of age. The primary hypotheses tested 1) the noninferiority of concomitant versus nonconcomitant vaccination with regard to Varicella zoster virus (VZV) Geometric Mean Titer (GMT) antibody responses, 2) the acceptability of geometric mean fold rise in VZV antibody response after concomitant vaccination, and 3) the noninferiority of concomitant versus nonconcomitant vaccination with regard to influenza virus strain-specific GMT antibody responses.

ELIGIBILITY:
Inclusion Criteria:

* Has history of varicella or residence in a VZV-endemic area for ≥30 years
* Is male, female not of reproductive potential, or female of reproductive potential and has a negative pregnancy test and agrees to avoid becoming pregnant throughout the study

Exclusion Criteria:

* Has history of hypersensitivity to any vaccine component
* Has previously received any varicella or zoster vaccine
* Has received an influenza vaccine for the 2015-16 season
* Has history of Herpes zoster
* Has received immunoglobulin, monoclonal antibodies, or any blood products within 5 months before study vaccination
* Is pregnant or breastfeeding, or expecting to conceive during the study
* Has used immunosuppressant therapy
* Has known or suspected immune dysfunction
* Has experienced Guillain-Barré syndrome within 6 weeks
* Has severe thrombocytopenia or any other coagulation disorder

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Levin MJ, Buchwald UK, Gardner J, Martin J, Stek JE, Brown E, Popmihajlov Z. Immunogenicity and safety of zoster vaccine live administered with quadrivalent influenza virus vaccine. Vaccine. 2018 Jan 2;36(1):179-185. doi: 10.1016/j.vaccine.2017.08.029. Epub 2017 Aug 19. PMID 28830693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 901 participants were screened and 882 were randomized to one of two vaccination groups.
Period: Overall Study
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Started | 441 (Participants are included as treated) | 441 (Participants are included as treated)
Vaccinated on Day 1 | 440 | 441
Vaccinated at Week 4 | 432 | 424
Completed | 438 | 437
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants are included as randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination | Total
Number analyzed (Participants) | 440 | 442 | 882
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (7.2) | 61.3 (7.7) | 61.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 262 | 528
  Male | 174 | 180 | 354

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Varicella-zoster Virus (VZV) Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Antibody
Description: Anti-VZV antibodies were determined using a Glycoprotein Enzyme-linked Immunosorbent Assay. Baseline was Day 1 for the Concomitant group and Week 4 for the Nonconcomitant group.
Time Frame: Baseline and 4 weeks after ZOSTAVAX™ vaccination (Week 4 for Concomitant group and Week 8 for Nonconcomitant group)
Population: Participants who met the inclusion criteria, were not protocol violators in a way that could influence the participant's immune response to study vaccine, received the quadrivalent influenza vaccine and ZOSTAVAX™ within the specified day ranges, and had samples for serology obtained within the specified day ranges.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 440 | 441
gpELISA units/mL
  Baseline, n=427, 409 | 206.0 [185.6 to 228.6] | 230.5 [208.4 to 255.0]
  Week 4, n=409, 392 | 395.6 [363.7 to 430.4] | 482.0 [446.4 to 520.4]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Nonconcomitant Vaccination; Test type: Non-Inferiority or Equivalence — A lower bound of the 95% CI on the fold difference (GMT ratio [Concomitant / Nonconcomitant] at 4 weeks postvaccination) >0.67 implied that the difference is statistically significantly noninferior to the prespecified clinically relevant decrease of 1.5-fold. A p-value ≤0.025 also supported a conclusion of noninferiority; p < 0.001, Longitudinal regression model; GMT ratio, 95% CI and p-value were based on a longitudinal regression model adjusting for prevaccination titers and age; GMT Ratio at 4 weeks postvaccination = 0.87, 95% CI 2-sided [0.80 to 0.95]

2. Primary Outcome: Geometric Mean Fold Rise From Baseline in VZV gpELISA Antibody Titers
Description: as for outcome 1
Time Frame: Baseline and 4 weeks after ZOSTAVAX™ vaccination (Week 4 for Concomitant group and Week 8 for Nonconcomitant group)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of titers (Week 4 / Baseline)
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 403 | 387
Ratio of titers (Week 4 / Baseline) | 1.9 [1.8 to 2.1] | 2.1 [1.9 to 2.2]
Statistical Analysis 1: Comparison: Concomitant Vaccination; Test type: Superiority or Other; p < 0.001, Longitudinal regression — A lower bound of the 95% CI on the GMFR > 1.4 indicated that the Concomitant Group induces an acceptable VZV antibody response. A p-value ≤0.025 also supported this conclusion; GMFR from Baseline = 1.90, 95% CI 2-sided [1.76 to 2.05] — Estimated GMFR, 95% CI and p-value were based on a longitudinal regression model adjusting for age

3. Primary Outcome: Geometric Mean Titers of H1N1-specific Influenza Virus Antibody
Description: Antibodies to H1N1-specific influenza virus hemagglutinin were measured using a Hemagglutinin Inhibition (HAI) assay. Antibody titers are the reciprocal of the highest dilution of serum that completely inhibited hemagglutinin.
Time Frame: Baseline and 4 weeks after Influenza vaccination (Week 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 440 | 441
Titer
  Baseline, n=426, 427 | 51.9 [45.4 to 59.3] | 50.1 [44.3 to 56.7]
  Week 4, n=409, 405 | 207.3 [185.6 to 231.7] | 200.5 [180.3 to 222.9]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Nonconcomitant Vaccination; Test type: Non-Inferiority or Equivalence — A lower bound of the 95% CI on the fold difference (GMT ratio [Concomitant / Nonconcomitant] at 4 weeks postvaccination) >0.67 implied that the difference is statistically significantly noninferior to the prespecified clinically relevant decrease of 1.5-fold. A p-value ≤0.025 also supported the conclusion of noninferiority; p < 0.001, Longitudinal regression; GMT ratio, 95% CI and p-value were based on a longitudinal regression model adjusting for prevaccination titers and age; GMT Ratio at 4 weeks postvaccination = 1.02, 95% CI 2-sided [0.88 to 1.18]

4. Primary Outcome: Geometric Mean Titers of H3N2-specific Influenza Virus Antibody
Description: Antibodies to H3N2-specific influenza virus hemagglutinin were measured using a Hemagglutinin Inhibition (HAI) assay. Antibody titers are the reciprocal of the highest dilution of serum that completely inhibited hemagglutinin.
Time Frame: Baseline and 4 weeks after Influenza vaccination (Week 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 440 | 441
Titer
  Baseline, n=426, 427 | 29.5 [26.2 to 33.3] | 31.1 [27.5 to 35.1]
  Week 4, n=409, 405 | 298.8 [264.1 to 338.1] | 272.0 [241.6 to 306.1]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Nonconcomitant Vaccination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, Longitudinal regression; GMT ratio, 95% CI and p-value were based on a longitudinal regression model adjusting for prevaccination titers and age; GMT Ratio at 4 weeks postvaccination = 1.10, 95% CI 2-sided [0.94 to 1.29]

5. Primary Outcome: Geometric Mean Titers of B-Yamagata-specific Influenza Virus Antibody
Description: Antibodies to B-Yamagata-specific influenza virus hemagglutinin were measured using a Hemagglutinin Inhibition (HAI) assay. Antibody titers are the reciprocal of the highest dilution of serum that completely inhibited hemagglutinin.
Time Frame: Baseline and 4 weeks after Influenza vaccination (Week 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 440 | 441
Titer
  Baseline, n=426, 427 | 14.6 [13.3 to 16.1] | 12.6 [11.6 to 13.7]
  Week 4, n=409, 405 | 46.7 [42.0 to 52.0] | 43.9 [39.7 to 48.6]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Nonconcomitant Vaccination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, Longitudinal regression; GMT ratio, 95% CI and p-value were based on a longitudinal regression model adjusting for prevaccination titers and age; GMT Ratio at 4 weeks postvaccination = 1.00, 95% CI 2-sided [0.88 to 1.14]

6. Primary Outcome: Geometric Mean Titers of B-Victoria-specific Influenza Virus Antibody
Description: Antibodies to B-Victoria-specific influenza virus hemagglutinin were measured using a Hemagglutinin Inhibition (HAI) assay. Antibody titers are the reciprocal of the highest dilution of serum that completely inhibited hemagglutinin.
Time Frame: Baseline and 4 weeks after Influenza vaccination (Week 4)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Number analyzed (Participants) | 440 | 441
Titer
  Baseline, n=426, 427 | 11.2 [10.3 to 12.2] | 10.4 [9.6 to 11.2]
  Week 4, n=409, 405 | 33.9 [30.5 to 37.7] | 32.3 [29.0 to 35.9]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Nonconcomitant Vaccination; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, Longitudinal regression; GMT ratio, 95% CI and p-value were based on a longitudinal regression model adjusting for prevaccination titers and age; GMT Ratio at 4 weeks postvaccination = 0.99, 95% CI 2-sided [0.87 to 1.13]

ADVERSE EVENTS:
Time Frame: Up to 28 days after any vaccination (up to Week 8)
Description: The population analyzed was all randomized participants who received at least one dose of study vaccination and had follow-up.
Arm/Group | Concomitant Vaccination | Nonconcomitant Vaccination
Serious Adverse Events (participants affected / at risk) | 4/435 | 6/438
Other Adverse Events (participants affected / at risk) | 256/435 | 256/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=435) | Nonconcomitant Vaccination (N=438)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteric cancer local (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=435) | Nonconcomitant Vaccination (N=438)
Injection site erythema (General disorders) | 153 (186) | 134 (150)
Injection site pain (General disorders) | 209 (322) | 211 (335)
Injection site pruritus (General disorders) | 33 (38) | 32 (33)
Injection site swelling (General disorders) | 102 (125) | 109 (125)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.